CLINICAL TRIAL: NCT05875155
Title: Ovarian Tissue Cryopreservation for Fertility Preservation in Patients Facing Infertility-causing Diseases or Treatment Regimens
Brief Title: Ovarian Tissue Cryopreservation for Fertility Preservation
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Other Study IDs: STUDY19080200
Record Dates: First submitted 2023-04-13; First posted 2023-05-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Autoimmune Diseases
Keywords: Fertility; Fertility Preservation; Infertility; Ovary; Ovarian; Oncofertility
MeSH Terms: conditions — Neoplasms; Autoimmune Diseases; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ovarian Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cryopreservation: Participants will have autologous ovarian tissue cryopreserved for fertility preservation.
  Interventions: Diagnostic Test: Infectious Disease Labwork; Diagnostic Test: Fertility-Based Labwork

INTERVENTIONS:
Diagnostic Test: Infectious Disease Labwork — Infectious disease labs will be drawn and resulted.
Diagnostic Test: Fertility-Based Labwork — Other labwork to understand fertility may be drawn.

SUMMARY:
The goal of this observational study is to learn about fertility preservation for pre-pubertal, peri-pubertal, and adult participants that are unable to pursue clinical standard of care fertility preservation such as egg (oocyte) and embryo cryopreservation.

In addition, this study will provide research tissue for the following Specific Aims:

1. To optimize techniques for cryopreservation of ovarian tissues from patients at significant risk for infertility.
2. To investigate factors affecting successful maturation ovarian tissue.

Participants will undergo a surgical procedure to remove an ovary (oophorectomy) to preserve their gonadal tissue for fertility preservation.

DETAILED DESCRIPTION:
The cure rate of cancer in children, adolescents and young adults continues to increase with advances in chemotherapy and/or radiation protocols. As more pediatric oncology patients become long-term survivors, the consequences of their treatment on their quality of life have become an important thrust of clinical oncology and basic science research. One of the most common and most devastating long-term sequelae following cancer treatment is infertility. Many chemotherapy and radiation-containing regimens for cancer therapy or prior to bone marrow transplantation can cause sterility in children and young adults. Fertility-preserving options are available for adult women (embryo freezing), but not all adult women are able to take advantage of this option since it requires fertilization. Some adult women are not able to cryopreserve embryos because they lack a partner or cannot delay treatment for the time required for ovarian stimulation. Currently, no fertility-preserving options are available for prepubescent girls who are not yet producing mature gametes and post-pubescent females whose follicular pool cannot be shielded from cancer therapy. However, experimental techniques are currently being developed to provide future alternatives for patients that preserve their ovarian tissue/cells prior to gonadotoxic treatment. In order to take advantage of these and future technologies, patients must harvest and preserve their ovarian tissue and/or oocytes (eggs) prior to the initiation of gonadotoxic therapy. This study will be available to girls and women from prepubertal years through 40 years of age who will undergo potentially sterilizing treatments. The primary objective of the proposed study is to develop techniques for long-term preservation of ovarian function through cryopreservation of ovarian tissue and/or cells prior to therapies that are likely to cause infertility (e.g., chemotherapy, radiation). This study will maintain cryopreserved ovarian tissue and/or cells for participating patients as a resource for future elective procedures to attempt fertility restoration. This study will also provide long-term follow-up on the fertility status of patients that will undergo a potentially sterilizing treatment for their primary disease or condition.

Fertility status has an important impact on the post-treatment quality of life for cancer survivors and other patients that receive gonadotoxic therapies (e.g., prior to bone marrow transplantation). Established fertility preserving therapies are available for adult women, but these therapies are not accessible or appropriate for all adult female patients. Currently there are no therapies to preserve the future fertility of preadolescent girls. However, new reproductive therapies are under development and may one day offer "fertile hope" to those survivors that do not currently have access to fertility preserving therapies. Clinical management of fertility-threatening diseases and treatments must have foresight of the gonadotoxic side effects and the potential for infertility. When no established fertility sparing options are available, it is reasonable to offer harvesting and cryopreservation of ovarian tissue as a possible means of fertility preservation. This study will provide a pool of research tissue that will be used to develop and test methods for manipulation and cryopreservation of ovarian tissue. Progress in these investigations may open up a range of new fertility preservation techniques to female patients that currently have no options. At the same time, a substantial portion of the patient's ovarian tissue will be cryopreserved and reserved for her own future use.

ELIGIBILITY:
Inclusion Criteria:

* Be female age less than 40 years old.
* Unable or unwilling to make use of oocyte or embryo banking alone.
* Be scheduled to undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy with risk of causing permanent and complete loss of subsequent ovarian function.
* Or, have a medical condition or malignancy that requires removal of all or part of one or both ovaries.
* Or, Have newly diagnosed or recurrent disease. Those who were not enrolled at the time of initial diagnosis (i.e., patients with recurrent disease) are eligible if they have not previously received therapy that is viewed as likely to result in complete and permanent loss of ovarian function.
* Have two ovaries if undergoing elective removal of an ovary for fertility preservation only.

Exclusion Criteria:

* Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
* Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.

Max Age: 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible patients who will undergo an infertility-causing treatment and for whom standard of care fertility preservation procedures are not available will be identified by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01-13 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Develop techniques for long-term preservation of female ovarian function through cryopreservation (freezing) of ovarian tissue and/or cells prior to therapies that are likely to cause infertility (e.g., chemotherapy, radiation). | [10 years]
  Treatment with specific chemotherapeutic agents and regimens induces prolonged absence of menstrual cycle in women of reproductive age. Sterilizing agents are thought to act directly on the ovary and produce premature ovarian insufficiency. Techniques will be developed through utilizing scientifically proven standards for long-term preservation of ovarian tissue and/or cells prior to gonadotoxic treatment.
Maintain cryopreserved ovarian tissue and/or cells for participating patients as a resource for future elective procedures to attempt fertility restoration. | [10 years]
  Ovarian tissue containing immature oocytes has been successfully cryopreserved in several animal models. When thawed, this tissue can be grafted into a host with resumption of both endocrine and reproductive function. Ovarian tissue cryopreservation has the important advantage of not requiring controlled ovarian hyperstimulation, thus, eliminating the delay in cancer therapy as well as elevated estradiol levels in patients with hormone sensitive cancers. After cancer therapy, participants can utilize their frozen ovarian tissue for transplantation or other applications, as eligible.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/ University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish individual participant data. The investigators will also report each individual participants data back to them. Participants will be identified with unique ID numbers. No identifiable information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: We will only share IPD with the patient (and only the patient) within one year of enrollment. We share study protocol and ICF with collaborating sites annually.
Access Criteria: De-identified research data will be shared with collaborators via a-mail, and with the broader scientific community via publication and presentations at national/international meetings.